CLINICAL TRIAL: NCT00159289
Title: Effect of Endotoxin on Inflammatory Markers in Exhaled Breath, Sputum, Saliva and Nasal Lavage in Healthy Non-Smokers and Current Smokers Including Patients With COPD
Brief Title: Endotoxin and Inflammatory Markers in Healthy Non-Smokers and Current Smokers Including Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No resources available
Sponsor: Imperial College London (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2002AT032B
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Mild to moderate Chronic Obstructive Pulmonary Disease (COPD); Volunteers (healthy non-smokers); Volunteers (current or ex-smokers)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Inhalation of LPS
  Interventions: Procedure: Inhalation of LPS
- 2 (Placebo Comparator): PLacebo
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Inhalation of LPS
  Arms: 1
Procedure: Placebo
  Arms: 2

SUMMARY:
The primary aim of this study is to investigate the effects of inhaled lipopolysaccharide endotoxin (LPS) on bronchial and alveolar exhaled nitric oxide (NO) and NO metabolites and other inflammatory markers and mediators in exhaled breath condensate, induced sputum, nasal lavage and mouthwash fluid in healthy non-smokers and current smokers, including patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smokers: normal spirometry (forced expiratory volume in 1 second [FEV1] more than or equal to 90% predicted) and normal exhaled NO (between 8 and 24 ppb; flow 50 ml/s)
* 0: At risk (current or ex-smokers): normal spirometry, with or without chronic symptoms (cough, sputum production)
* I-II: Mild-moderate COPD

  * FEV1 reversibility of < 15% after inhaled beta2-agonists
  * FEV1/forced vital capacity (FVC) < 70% predicted
  * FEV1 between greater than or equal to 50% and less than 80%
  * With or without chronic symptoms (cough, sputum production)
* Able to comprehend and grant a written informed consent

Exclusion Criteria:

* Concomitant use or pre-treatment within the last 4 weeks with oral steroids
* Respiratory infection within 4 weeks prior to entry into the trial
* Females who are pregnant or lactating
* History of current or past drug or alcohol abuse

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
sputum induced

CONTACTS AND LOCATIONS:
Overall Officials: Sergei A Kharitonov, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Section of Airway Disease, Asthma Lab, Imperial College London, Royal Brompton Hospital, London, United Kingdom